CLINICAL TRIAL: NCT02275949
Title: The Efficacy and Safety of Acupuncture for Cerebral Vasospasm After Subarachnoid Hemorrhage
Brief Title: Acupuncture for Cerebral Vasospasm After Subarachnoid Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Seong-Uk Park, A full professor, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACUSAH20141059
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: SAH (Subarachnoid Hemorrhage); Cerebral Vasospasm
Keywords: SAH (Subarachnoid Hemorrhage); Cerebral Vasospasm; Acupuncture
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — Acupuncture Therapy; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Experimental): acupuncture, electroacupuncture and intradermal acupuncture are done at every session.
  Interventions: Device: acupuncture; Device: Electroacupuncture; Device: Intradermal acupuncture
- Control group (Sham Comparator): Mock transcutaneous electrical nerve stimulation(mock TENS) and sham intradermal acupuncture are carried out.
  Interventions: Device: Mock transcutaneous electrical nerve stimulation; Device: sham intradermal acupuncture

INTERVENTIONS:
Device: acupuncture — Acupuncture needles are inserted at the acupoints Zusanli(ST 36), Neiguan(PC 6), Gongsun(SP 4), and Xiangu(ST 43) bilaterally.
  Arms: Study group
Device: Electroacupuncture — The electric stimulator will be connected to the handles of each needles on the ST 36 and PC 6 bilaterally with 5Hz.
  Arms: Study group
Device: Intradermal acupuncture — Intradermal acupuncture needles with tape are inserted on the ST36, PC6, SP4, ST43 bilaterally and maintained until the next session.
  Arms: Study group
Device: Mock transcutaneous electrical nerve stimulation — Electrical insulator are attached on the ST36 and PC6 bilaterally, the same electric stimulator will be connected on the points with the same parameters as the study group, but without current intensity.
  Other Names: Mock TENS
  Arms: Control group
Device: sham intradermal acupuncture — Intradermal acupuncture needles are put over the tape not penetrating the skin.
  Arms: Control group

SUMMARY:
This study will evaluate acupuncture's effect of preventing vasospasm after SAH.

A total of 80 participants will be recruited and will be randomized to a study group or a control group. Acupuncture, electroacupuncture and intradermal acupuncture will be done at every session in a study group, while mock transcutaneous electrical nerve stimulation(mock TENS) and sham intradermal acupuncture will be carried out in a control group.

DETAILED DESCRIPTION:
Intervention starts within 96hours after SAH, after ruptured aneurysms have been secured by endovascular coiling or surgical clipping. Intervention is applied once a day, 6 days a week for 2 weeks(total 12 sessions) in addition to standard treatment such as prophylactic HHH therapy and nimodipine. Sterile disposable, stainless steel acupuncture needles are used.

Primary outcome measurement is the occurrence of delayed ischemic neurological deficit between the study group and the control group. Moreover, the incidence of angiographic vasospasm, TCD vasospasm, and vasospasm-related infarct on CT or MRI, the change of nitric oxide(NO) and endothelin-1 in plasma, mortality and participant's functional status using mRS will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Participants conforming to all the following conditions will be included: 1) SAH verified by CT and cerebral angiography; 2) aneurysm treated by endovascular coiling or surgical clipping; 3) age > 18 years; 4) HHS 1-4; 5) acupuncture treatment can start within 96 hours after SAH; 6) participation is voluntarily and the informed consent signed.
* Healthy controls who matched with patients in gender and age

Exclusion Criteria:

* Participants with any of the following conditions will be excluded: 1) traumatic or infectious SAH; 2) HHS 5; 3) Transcranial Doppler (TCD) cannot performed; 4) heart, liver or renal failure; 5) presence of cardiac pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The occurrence of delayed ischemic neurological deficit | 14 days
  The occurrence of delayed ischemic neurological deficit between the study group and the control group will be compared. DIND is defined as an unaccountable new focal neurological deficit lasting more than 2hours. Any occurrence of DIND will be recorded by the physician and verified by the investigator every day.

SECONDARY OUTCOMES:
The incidence of angiographic vasospasm | 14 days
  Angiographic vasospasm is defined as focal or generalized reduction of cerebral arterial caliber on conventional cerebral angiogram or computed tomographic angiography confirmed by a neuroradiologist and neurosurgeon.
The incidence of TCD vasospasm | 14 days
  TCD vasospasm is defined as Peak systolic middle cerebral artery velocity > 200cm/s and Lindegaard ratio >3
The incidence of vasospasm-related infarct on CT or MRI | 14 days
  It is defined as cerebral infarction in the region of angiographic vasospasm or TCD vasospasm is shown on CT or MRI
The change of nitric oxide(NO) and endothelin-1 in plasma | 14days
  Blood sample of 3ml is taken from brachial vein and centrifuged by 3000 rpm for 15minutes and kept in a freezer before analysis. Blood sample will be taken twice, before the start of treatment and after the end of treatment. In addition, the level of serum NO and endothelin-1 between patients and healthy controls will be compared.
Mortality | 14 days and 28 days
  Mortality at the end of treatment and 14days after the treatment(or at discharge)
modified Rankin Scale (mRS) | 14 days and 28 days
  The participan's functional status at the end of treatment and 14days after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Uk Park, KMD, PhD, Principal Investigator — Stroke & Neurological Disorders Center, Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, Gangdong-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei JJ, Guo RJ, Fu GJ, Liang X, Xu ZM, Jia M, Zeng ZX, Du WQ, Jiao WW, Sun LJ, Liu HM, Guo CL, Tong CG, Zhang YL, Liao X. Registration of intervention trials of Traditional Chinese Medicine for four neurological diseases on Chinese Clinical Trial Registry and ClinicalTrials.gov: a narrative review. J Tradit Chin Med. 2022 Feb;42(1):148-153. doi: 10.19852/j.cnki.jtcm.2022.01.010. PMID 35294135
- [Derived] Lee DH, Cho SY, Yang SB, Lee HM, Shin HS, Lee SH, Koh JS, Kwon S, Jung WS, Moon SK, Park JM, Ko CN, Kim H, Park SU. Efficacy of Acupuncture Treatment to Prevent Cerebral Vasospasm After Subarachnoid Hemorrhage: A Double-Blind, Randomized Placebo-Controlled Trial. J Altern Complement Med. 2020 Dec;26(12):1182-1189. doi: 10.1089/acm.2020.0156. Epub 2020 Sep 1. PMID 32876468
- [Derived] Cho SY, Lee DH, Shin HS, Lee SH, Koh JS, Jung WS, Moon SK, Park JM, Ko CN, Kim H, Park SU. The efficacy and safety of acupuncture for cerebral vasospasm after subarachnoid hemorrhage: study protocol for a randomized controlled trial. Trials. 2015 Feb 28;16:68. doi: 10.1186/s13063-015-0591-7. PMID 25886483